CLINICAL TRIAL: NCT06207006
Title: Conquering Fear Online: a Pilot Randomised Controlled Trial Assessing the Efficacy and Feasibility of an Internet-based Self-management Intervention on Subclinical Fear of Cancer Recurrence
Brief Title: E-intervention on Subclinical Fear of Cancer Recurrence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW22-602
Record Dates: First submitted 2023-12-12; First posted 2024-01-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Cancer; Psychooncology; Fear of Cancer Recurrence
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective, parallel RCT design will be used to assess the impact of the eConquerFear-HK intervention on FCR improvement among Chinese cancer survivors in Hong Kong. Participants will be randomly assigned to an intervention group or a control group at a 1:1 ratio, using a computer-generated block randomization sequence generated by a statistician who is blinded to the identity of participants. This allocation concealment approach minimizes risk of selection and assessment bias. The serially labelled opaque sealed envelope method will be used for randomization. Block randomization structure with randomly permuted blocks sizes of 2 and 4 will be used to ensure close balance of numbers in each arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to the intervention or control arms.
  The participants are masked in terms of not knowing that the intervention, eConquerFear-HK are hypothesized to yield larger effects than the other (i.e. control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- eConquerFear-HK (Experimental): Participants in the eConquerFear-HK intervention group will receive six online modules with each containing educational text, illustrative graphics, interactive exercises, and brief videos. Every module will teach a specific topic, such as self-examination and medical surveillance, values-based goal setting, attention training, detached mindfulness, worry management and treatment summary and relapse prevention.
  Interventions: Behavioral: eConquerFear-HK
- Basic Cancer Care (Active Comparator): Participants in the control group will receive six videos, which were designed to provide comprehensive lifestyle guidance (e.g., relaxation techniques, diet and physical activity advices) to help with survivors' maintenance of health in long-term.
  Interventions: Behavioral: Basic Cancer Care

INTERVENTIONS:
Behavioral: eConquerFear-HK — The key goals of the intervention are to: (i) teach strategies for controlling worry and excessive threat monitoring; (ii) modify underlying unhelpful MCQ beliefs about worry; (iii) develop appropriate monitoring and screening behaviours, (iv) encourage acceptance of the uncertainty brought about by a cancer diagnosis, and (v) clarify values and encourage engagement in values-based goal setting.
  Arms: eConquerFear-HK
Behavioral: Basic Cancer Care — Basic Cancer Care serves as an active comparator and is not developed specifically to target fear of cancer recurrence through modifying participants' cognitive beliefs. Participants in this arm will receive 6 videos about relaxation, generic dietary and exercise knowledge.
  Arms: Basic Cancer Care

SUMMARY:
The present study aims to adapt a metacognition-based ConquerFear-HK to an internet-based self-management intervention, namely eConquerFear-HK and evaluate in a randomised controlled trial, its feasibility, utility, and potential effectiveness on fear of cancer recurrence reduction among local Chinese cancer survivors with subclinical fear of cancer recurrence.

DETAILED DESCRIPTION:
A pilot randomised controlled feasibility trial will used to test the feasibility, utility, and potential effectiveness of an internet-based self-management intervention for fear of cancer recurrence among local Chinese cancer survivors with subclinical fear of cancer recurrence.

The following hypotheses will be tested:

1. There will be a greater FCR improvement in cancer survivors receiving eConquerFear-HK intervention vs those in the active control group.
2. There will be a greater MCQ reduction in cancer survivors receiving eConquerFear-HK intervention vs those in the active control group.
3. There will be greater improvements in secondary outcomes (psychological distress and quality of life) in cancer survivors receiving eConquerFear-HK intervention vs those in the active control group.
4. Cancer survivors receiving eConquerFear-HK intervention will perceive the intervention useful for managing their FCR and be satisfied with the intervention.
5. Cancer survivors receiving eConquerFear-HK intervention will show high completion rates.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese- or Mandarin-speaking Chinese cancer survivors
* recently diagnosed with potentially curable (stage 0 to III) colorectal or breast cancer
* had recently completed surgery as primary treatment
* have completed hospital-based adjuvant treatments (including radiotherapy and chemotherapy) within the past six months
* scored 13 to 21 on the fear of cancer recurrence-short form will be recruited.

Exclusion Criteria:

* non-Chinese ethnicity
* metastatic cancer
* with current diagnosis of depression or psychosis or are currently receiving psychological treatments
* language or intellectual difficulties that prevent them from understanding the intervention content
* having limited or no Internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of subject recruitment | baseline
  number of participants consent and being randomized/number of eligible patients x 100
Rate of subject retention | baseline,3-months post-intervention and 6-months post-intervention
  number of participants who complete follow-up assessments at 3 and 6 months post-baseline/number of participants enrolled x 100
Adherence rate to intervention | the immediate post-intervention
  number of participants who complete the intervention/number of being allocated to attend the intervention x 100
Intervention utility | the immediate post-intervention
  Intervention utility will be assessed using the site use metrics, including total number of log-ins
Acceptability of the intervention | the immediate post-intervention
  Acceptability of the intervention will be assessed using the 22-item measure, which was adopted from the 31-item measure designed to assess the general views on the presentation and content of information in a decision aid intervention for treatment decision making. It assess the comprehensibility of the intervention content and also its utility using 4- (1 = "Poor"; 2 = "Fair"; 3 = "Good"; 4 = "Excellent") or 5-option (1 ="strongly disagree"; 5 = "strongly agree") categorical responses, respectively. Higher scores indicate better acceptability.
Change of fear of cancer recurrence | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  Fear of cancer recurrence. FCR will be assessed using the Chinese 42-item Fear of Cancer Recurrence Inventory (FCRI) at four assessment points (T0-T3).(5) FCRI comprises seven subscales: trigger, severity, psychological distress, functional impairment, reassurance, insights and coping strategies measured using 5-point Likert scales (0 = "never"; 4 = " a great deal or all the time").(5) Total scores range from 0 to 168; with higher scores indicating higher FCR.

SECONDARY OUTCOMES:
Change of quality of life | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  Quality of life will be measured by the Chinese version of the 30-item European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30), consisting of five functional subscales (physical, role, emotional, cognitive, and social functioning), three symptom subscales (pain, fatigue and nausea/vomiting), a global health subscale, five single symptom items (e.g., sleep disturbance, dyspnea, appetite loss, constipation, and diarrhea), and an single item for financial difficulty. The score range is 0-100. High scores on the functional and global health subscales indicate better functioning and QoL, respectively. High scores on the symptom subscale or item indicate more symptom(s).
Change of general psychological distress | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  e Chinese 14-item Hospital Anxiety and Depression Scale (HADS),(21) comprising two 7-item subscales that measure anxiety and depression. Each subscale total scores range from 0 to 21 with higher scores suggesting higher distress.
Attitude towards internet assessed using categorical Likert scales | the immediate post-intervention
  Attitude towards internet will be assessed using a 6 points-categorical Likert scale (0-5) asking if they find internet easy to use. Higher scores indicate more positive attitude towards internet.
Treatment satisfaction | the immediate post-intervention
  A 17-item treatment satisfaction questionnaire, originally designed to evaluate overall satisfaction with the intervention in our current RCT of ConquerFear-HK, will be used. The first 9 items will be assessed using a 5 points-categorical Likert scale (1-5) Higher scores indicate higher satisfaction. The remaining questions are open-questions.
Change of metacognition | Baseline, the immediate post-intervention, 3-months post-intervention and 6-months post-intervention
  Metacognition will be assessed at T0-T3 using the 30-item Metacognitions Questionnaire- 30 (MCQ-30), consisting of five subscales assessing Positive beliefs about worry, Negative beliefs about worry, Cognitive Self-Consciousness, Cognitive Confidence, and Need to control thoughts. A 4 points-categorical Likert scale (1-4) will be used. Higher scores indicate worse metacognition

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Ng, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- Queen Mary Hospital-Department of Surgery, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.